CLINICAL TRIAL: NCT05810844
Title: Comparison Of Effects of Motor Relearning Program (MRP) Versus Neuro Development Treatment (NDT) For Balance and Gait in Chronic Ischemic Stroke Patients: A Randomized Clinical Trial
Brief Title: Comparison Of Effects of MRP Vs NDT For Balance and Gait in Chronic Ischemic Stroke Patients RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/522
Record Dates: First submitted 2023-03-15; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Relearning Program (MRP) (Experimental)
  Interventions: Diagnostic Test: Motor Relearning Program (MRP)
- Neuro Development Treatment (NDT) (Experimental)
  Interventions: Diagnostic Test: Neuro Development Treatment (NDT)

INTERVENTIONS:
Diagnostic Test: Motor Relearning Program (MRP) — MRP technique with a conventional physiotherapy treatment. Conventional physiotherapy treatment will help to reduce the functional impairments in chronic ischemic stroke
  Arms: Motor Relearning Program (MRP)
Diagnostic Test: Neuro Development Treatment (NDT) — Neuro-Development Treatment NDT as well as conventional treatment. Conventional physiotherapy treatment will help to reduce the functional impairments in chronic ischemic stroke patients
  Arms: Neuro Development Treatment (NDT)

SUMMARY:
To determine the comparison between effects of Motor Relearning Program (MRP) and Neuro-Development Treatment (NDT) on balance and gait in chronic ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic ischemic stroke Patients more than 6 months. (55)
2. Patient with good cognitive status minimum 20 or greater out of 30 in Mini mental state examinations.(56)
3. Age between 45-65 years.(57)
4. Patient with limb spasticity equal to 2 or less than 2 on Modified Ashworth scale.(56)
5. Both male and female patients.(58)

Exclusion Criteria:

1. History of neurologic disease(59, 60)
2. History of lower limb fracture.(61)
3. History of spinal cord fracture.(61)
4. Patient with skin discoloration, skin ulcers and skin allergy.(62)
5. Patients with a history of the recurrent stroke. (63)
6. Patients with any peripheral vascular disease.(60)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Effects of Motor Relearning Program Techinique, Neuro Development Treatment Techinique | 6 Months

IPD SHARING:
Plan to Share IPD: No